CLINICAL TRIAL: NCT01945229
Title: Thumb-ECG Ambulant Screening for Atrial Fibrillation in Patients Treated for Hyperthyroidism (TAMBOURINE)
Acronym: TAMBOURINE
Status: Terminated | Type: Observational
Why Stopped: Preliminary analyses of data indicated study should be terminated for futility
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Peter Giesecke, M.D, M.D., specialist internal medicine and cardiology, Karolinska Institutet
Other Study IDs: 3/9 B
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Hyperthyroidism; Atrial Fibrillation
MeSH Terms: conditions — Hyperthyroidism; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hyperthyroid patients: Patients with hyperthyroidism admitted for treatment with radioiodine or antithyroid drugs

SUMMARY:
Background: Atrial fibrillation is a common heart rhythm disturbance affecting some 1-2% of the western population. It may cause symptoms such as irregular heartbeats, shortness of breath, and fatigue. It may also be asymptomatic (ie "silent atrial fibrillation). In some cases, atrial fibrillation is permanent whereas in others it is sporadic. Regardless of symptoms, there is an increased risk of stroke in some patients with this condition. Novel technologies are being developed to increase detection of silent atrial fibrillation, in order to find patients who might benefit from treatment with oral anticoagulants (blood-thinning medications) in order to reduce the risk of stroke. One of these technologies is thumb-ECG, a simple way for a patient to have his or her heart rhythm reliably analyzed at home.

Hyperthyroidism (sometimes referred to as "toxic goiter") is defined as an excessive production of thyroid hormone. It is known that hyperthyroidism may cause atrial fibrillation in about 8% of cases.

Objective: To provide thumb-ECG-monitors to hyperthyroid patients before and after treating their hormonal disturbance, in order to find episodes of silent atrial fibrillation.

Design: Prospective observational study.

Hypotheses:

* Primary hypothesis: Silent atrial fibrillation is at least as common as overt atrial fibrillation in hyperthyroid patients.
* Secondary hypothesis nr 1: Atrial fibrillation continues to be more prevalent compared to the normal population even after hyperthyroidism is treated.
* Secondary hypothesis nr 2: The majority of patients with hyperthyroidism and atrial fibrillation are at increased risk of stroke and should be considered for treatment with oral anticoagulants.

ELIGIBILITY:
Inclusion Criteria:

* Patient is deemed suitable for treatment with radioiodine or antithyroid drugs
* Patient has a thyreotropin (TSH) value below 0,1 mIU/L, measured less than 2 weeks before inclusion
* Patient has a CHADS-VASc-score of 1 point or higher (excluding if 1 point is for female sex only)
* Patient gives written consent to participate in study

Exclusion Criteria:

* Patient has a previously known diagnosis of atrial fibrillation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will screen all patients residing in the extended region around Stockholm, Sweden who have been referred and admitted to the Radiumhemmet clinic for investigation (and usually treatment) with radioiodine. As of February 2016, we will also include patients referred for treatment with antithyroid drugs at the endocrinology clinics of 1) Sahlgrenska University Hospital, Gothemburg Sweden, 2) Karolinska University Hospital, Stockholm, Sweden, 3) Danderyds Hospital, Stockholm, Sweden
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2014-02; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Prevalence of asymptomatic (silent) atrial fibrillation in hyperthyroid patients | Upon inclusion and 2 weeks onwards
  Upon inclusion, each patient will receive a thumb-ECG-monitor to take home. He/she will register his/her heart rhythm twice daily, and can also register at will upon symptoms. This will continue for 2 weeks, after which the monitor is returned.

SECONDARY OUTCOMES:
Prevalence of asymptomatic (silent) atrial fibrillation in patients treated for hyperthyroidism. | Between 12 and 14 weeks after inclusion
  When a patient comes back to the policlinic after hyperthyroidism treatment (typically 3 months later), the same procedure is performed as upon inclusion. Thumb-ECG-monitoring is performed during a 2-week period.
Prevalence of risk factors for stroke in patients with atrial fibrillation | Momentary (day 1, upon inclusion)
  Risk factors for stroke in atrial fibrillation according to the CHADS-VASc-scoring system.

CONTACTS AND LOCATIONS:
Overall Officials: Mårten Rosenqvist, Prof, Study Chair — Karolinska Institutet
Locations (3):
- Sweden (3):
  - Medicine Clinic, Sahlgrenska University Hospital, Gothemburg
  - Endocrinology Clinik, Karolinska University Hospital, Stockholm
  - Medicine Clinic, Danderyds Hospital, Stockholm

REFERENCES:
- [Background] Frost L, Vestergaard P, Mosekilde L. Hyperthyroidism and risk of atrial fibrillation or flutter: a population-based study. Arch Intern Med. 2004 Aug 9-23;164(15):1675-8. doi: 10.1001/archinte.164.15.1675. PMID 15302638
- [Background] Osman F, Franklyn JA, Holder RL, Sheppard MC, Gammage MD. Cardiovascular manifestations of hyperthyroidism before and after antithyroid therapy: a matched case-control study. J Am Coll Cardiol. 2007 Jan 2;49(1):71-81. doi: 10.1016/j.jacc.2006.08.042. Epub 2006 Dec 13. PMID 17207725
- [Background] Metso S, Auvinen A, Salmi J, Huhtala H, Jaatinen P. Increased long-term cardiovascular morbidity among patients treated with radioactive iodine for hyperthyroidism. Clin Endocrinol (Oxf). 2008 Mar;68(3):450-7. doi: 10.1111/j.1365-2265.2007.03064.x. Epub 2007 Oct 17. PMID 17941909
- [Background] Camm AJ, Lip GY, De Caterina R, Savelieva I, Atar D, Hohnloser SH, Hindricks G, Kirchhof P; ESC Committee for Practice Guidelines (CPG). 2012 focused update of the ESC Guidelines for the management of atrial fibrillation: an update of the 2010 ESC Guidelines for the management of atrial fibrillation. Developed with the special contribution of the European Heart Rhythm Association. Eur Heart J. 2012 Nov;33(21):2719-47. doi: 10.1093/eurheartj/ehs253. Epub 2012 Aug 24. No abstract available. PMID 22922413